CLINICAL TRIAL: NCT01534260
Title: Phase I/II Study of Combination of Sorafenib, Vorinostat, and Bortezomib for the Treatment of Acute Myeloid Leukemia With Complex- or Poor-risk (Monosomy 5/7) Cytogenetics or FLT3-ITD Positive Genotype
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hamid Sayar (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Bayer (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Hamid Sayar, Assistant Professor of Clinical Medicine, Indiana University
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUCRO-0327; 1110007281 (Other: Indiana University IRB)
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Results first posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-07

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Sorafenib; Vorinostat; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- sorafenib, vorinostat and bortezomib (Experimental): Escalating cohorts of sorafenib, vorinostat and bortezomib
  Interventions: Drug: sorafenib, vorinostat and bortezomib

INTERVENTIONS:
Drug: sorafenib, vorinostat and bortezomib — Escalating dose cohorts of sorafenib, vorinostat and bortezomib. The first cohort will receive sorafenib from day 1 to 14, vorinostat will be given on days 1-4 and 8-12, and bortezomib will be given on days 1 and 8. This will be followed by 7 days of rest. Therefore each cycle will be 21 days.

SUMMARY:
This research is being done because treatment options are very limited and usually unsuccessful for Acute Myeloid Leukemia (AML) in older individuals, or younger people with disease that has relapsed and/or proven resistant to standard therapy. Subjects are invited to participate in this study that will examine the use of three drugs called Sorafenib (Nexavar), Vorinostat (Zolinza) and Bortezomib (Velcade) for treating acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed baseline diagnosis of AML by the revised guidelines of the International Working Group for AML including newly diagnosed, relapsed or refractory disease.
* Poor-risk or complex cytogenetics profile, or deletion of chromosome 5, or deletion of chromosome 7, or positive FLT3-ITD mutation.
* The patient must have discontinued all previous therapies for acute leukemia for at least 14 days and recovered from the acute non-hematologic side effects of the therapy.
* Hydroxyurea to control peripheral blood blast count must be discontinued within 24 hours prior to the initiation of treatment.
* Patients must have an ECOG (Zubrod) performance status of 0-2
* Patients must have adequate hepatic and renal function according to the protocol within one week prior to treatment.
* Female patients must be postmenopausal, surgically sterile or agree to use effective methods of contraception throughout the study.
* Male patients, even if surgically sterilized, must agree to practice effective contraception throughout the study.
* Patients must be able to swallow and tolerate oral medications.

Exclusion Criteria:

* Known central nervous system (CNS) leukemia.
* Diagnosis of acute promyelocytic leukemia (APL).
* Grade >/= 2 peripheral neuropathy.
* Serious illness including, significant ongoing or active infection, New York Heart Association (NYHA) Grade III or IV congestive heart failure, unstable angina or new onset angina or myocardial infarction within the past 6 months, cardiac ventricular arrhythmias requiring anti-arrhythmic therapy, thrombotic or embolic events such as a cerebrovascular accident including transient ischemic attacks within past 3 months. Serious medical or psychiatric illness/social situations that in the opinion of the investigator would limit compliance with study requirements.
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Active corneal erosions or history of abnormal corneal sensitivity test.
* Known or suspected history of severe hypersensitivity reaction to tyrosine kinase inhibitors, histone deacetylase inhibitors, proteosome inhibitors, boron, or mannitol.
* Female patients who are lactating or have a positive serum pregnancy test within 72 hours of initiation of treatment, or a positive urine pregnancy test on Day 1 before first dose of study drug.
* Concurrent use of other histone deacetylase inhibitors (e.g. valproic acid) are prohibited except for HDAC inhibitors or HDAC-inhibitor like agents used for non-cancer treatment (e.g. epilepsy), where a 14 day washout is allowed.
* Radiation therapy within 3 weeks before randomization.
* Patients with known HIV, or known active hepatitis B or C infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-02-10 (Actual); Primary Completion 2016-08-29 (Actual); Study Completion 2017-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Sayar, MD, Principal Investigator — Indiana University Melvin and Bren Simon Cancer Center
Locations (1):
- Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This protocol was based on enrolling up to 44 patients with 2 to 30 patients in phase I and 14 patients in phase II. The study enrolled 37 patients with 17 in phase I and 20 in phase II.
Groups:
- Phase I Dose Escalating: escalating dose cohorts of sorafenib, vorinostat and bortezomib. All cohorts will receive sorafenib from day 1 to 14 and vorinostat from day 1 to 4 and day 8 to 12. Bortezomib will be given on days 1 and 8 for all cohorts, with cohorts 4 and 5 also receiving bortezomib on days 4 and 11 for cycles 1 through 4. This will be followed by 7 days of rest. Therefore each cycle will be 21 days.
- Phase II at MTD: patients received sorafenib at 400 mg bid from day 1 to 14 and vorinostat 200 mg bid from day 1 to 14. Bortezomib will be given at 1.3 mg/m2 on days 1, 4, 8 and 11 for cycles 1-4, and then on days 1 and 8 for cycle 5 and beyond. Bortezomib will be given on days 1 and 8 beyond 4 cycles to reduce the risk of neurotoxicity.
Period: Overall Study
Arm/Group | Phase I Dose Escalating | Phase II at MTD
Started | 17 | 20
Completed | 1 | 0
Not Completed | 16 | 20
Not completed — Adverse Event | 1 | 8
Not completed — Death | 2 | 0
Not completed — Lack of Efficacy | 1 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Disease Progression | 8 | 6
Not completed — Physician Decision | 3 | 1
Not completed — No treatment, per protocol | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Escalating | Phase II at MTD | Total
Number analyzed (Participants) | 17 | 20 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 12 | 26
  >=65 years | 3 | 8 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (14.2) | 58.2 (14.8) | 55.2 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 18 | 35
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 14 | 19 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose Limiting Toxicity
Description: The number of patients who had a DLT during the dose finding/confirming portion (Phase I) of the trial for the safety of the combination of sorafenib, vorinostat, and bortezomib.
Time Frame: up to 9 months
Population: All Phase I patients receiving at least one dose of study drug and having at least one evaluable post-baseline visit
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Escalating
Number analyzed (Participants) | 17
Participants | 0

2. Primary Outcome: Phase II - Percentage of Patients With a Partial Response or Greater
Description: Evaluate the overall response rate of patients receiving therapy. Patients are considered as having a response if their overall response is Partial Response or better. The percentage of patients achieving this and the exact 95% confidence interval will be calculated. Responses will be defined using the response criteria determined by the International Working Group for AML.
Time Frame: up to 9 months
Population: All Phase II patients who received at least one dose of study drug and had at least one evaluable post-baseline visit
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II at MTD
Number analyzed (Participants) | 15
percentage of participants | 40.0 [16.3 to 67.7]

3. Secondary Outcome: Phase II - Time to Relapse
Description: Will be examined using Kaplan-Meier estimates. Time from date of confirmed complete remission to date of relapse. The observations of patients who died or remained alive and relapse free were censored at date of death or last disease evaluation, respectively.
Time Frame: Up to one year
Population: All Phase II patients who received at least one dose of study drug, had at least one evaluable post-baseline visit, and achieved complete remission
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase II at MTD
Number analyzed (Participants) | 3
days | 32 [22 to 42]

4. Secondary Outcome: Phase II - Treatment-Related Adverse Events Grade 3 or Higher
Description: Number of unique patients who had a treatment-related (possible, probable or definite) adverse events that were graded 3 or higher.
Time Frame: Up to one year
Population: All Phase II patients who received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II at MTD
Number analyzed (Participants) | 20
Participants | 4

ADVERSE EVENTS:
Time Frame: Up to one year
Arm/Group | Phase I Dose Escalating | Phase II at MTD
Serious Adverse Events (participants affected / at risk) | 7/17 | 11/20
Other Adverse Events (participants affected / at risk) | 16/17 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Escalating (N=17) | Phase II at MTD (N=20)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Eye disorders - Other (Eye disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 3 | 2
Lung infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 2
Neutrophil count decreased (Investigations) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Escalating (N=17) | Phase II at MTD (N=20)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Spleen disorder (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac disorders - Other (Cardiac disorders) | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 2
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Endocrine disorders - Other (Endocrine disorders) | 1 | 0
Eye disorders - Other (Eye disorders) | 0 | 2
Scleral disorder (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 4
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 5
Diarrhea (Gastrointestinal disorders) | 11 | 12
Dry mouth (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 2
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 2
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 6 | 5
Nausea (Gastrointestinal disorders) | 7 | 12
Oral hemorrhage (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 5 | 10
Edema face (General disorders) | 0 | 1
Edema limbs (General disorders) | 1 | 2
Fatigue (General disorders) | 2 | 3
Fever (General disorders) | 2 | 4
General disorders and administration site conditions - Other (General disorders) | 4 | 1
Hypothermia (General disorders) | 1 | 0
Localized edema (General disorders) | 2 | 1
Malaise (General disorders) | 1 | 0
Pain (General disorders) | 4 | 2
Allergic reaction (Immune system disorders) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Infections and infestations - Other (Infections and infestations) | 0 | 2
Papulopustular rash (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 2
Bruising (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Intestinal stoma site bleeding (Injury, poisoning and procedural complications) | 0 | 1
INR increased (Investigations) | 0 | 1
Urine output decreased (Investigations) | 1 | 0
Weight gain (Investigations) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 6 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 3
Hyponatremia (Metabolism and nutrition disorders) | 2 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 4
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 2
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Erythroderma (Skin and subcutaneous tissue disorders) | 2 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 3
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Hot flashes (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 3
Hypotension (Vascular disorders) | 4 | 2
Superficial thrombophlebitis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes